CLINICAL TRIAL: NCT06566105
Title: The Liver BIoBank Lombardia Genomic Cohort Study (LIVER-BIBLE): Personalized Medicine for the Management of Hepatic and Cardiovascular Thrombotic Complications of Fatty Liver
Brief Title: The Liver BIoBank Lombardia of Fatty Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Clinical Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LIVER BIBLE
Record Dates: First submitted 2024-03-07; First posted 2024-08-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: NAFLD; Precision Medicine; Cardiovascular Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROCEDURES RELATED TO THE STUDY (Other): * Selection of blood donors at risk of NAFLD and metabolic diseases and sample collection blood
  * Evaluation of early cardiovascular damage and characterization of liver damage in patients with high probability of severe NAFLD
  * Study of genomics and biomarkers
  * Generation of an in vitro genetic model of NAFLD
  Interventions: Genetic: precision medicine approach

INTERVENTIONS:
Genetic: precision medicine approach — precision medicine approach to improvement of risk stratification of hepatic and cardiovascular complications in non-alcoholic fatty liver disease in a group of healthy subjects at increased risk of metabolic pathologies

SUMMARY:
NAFLD is most frequently linked to excess adiposity, insulin resistance and cardiometabolic risk factors, it has become the leading cause of liver disease worldwide, and is associated with increased mortality due to multiple causes. HFC has a strong genetic component and the investigators recently showed that it plays a causal role in determining progressive liver disease and insulin resistance.

The genetic risk score predicting liver fat content (HFC-GRS) improves the stratification of liver related events, and the investigators have preliminary data on new common and rare variants that contribute to NAFLD susceptibility, and on a new non-invasive circulating biomarker associated with hepatic fat and lipotoxicity (Interleukin-32). However, no data are yet available on the causal role of hepatic fat on the procoagulant state associated with NAFLD, which could participate to liver damage and is a causal factor in atherothrombotic complications. The aim of the study is to examine the potential application of a precision medicine approach to the improvement of stratification of the risk of liver-related and cardiovascular thrombotic complications of hepatic fat accumulation (HFC) and non-alcoholic fatty liver disease (NAFLD), with a special focus on the role of procoagulant imbalance in mediating the at-risk phenotypes.

DETAILED DESCRIPTION:
The aims of the project will be:

* To examine whether a comprehensive HFC-GRS coupled with evaluation of environmental triggers, imaging techniques and novel circulating biomarkers help in stratifying of the risk of NAFLD and associated complications in a cohort of asymptomatic individuals at high risk from the general population (the Liver-Bible cohort). The Liver-Bible cohort is made up of >2,500 individuals with multiple metabolic risk factors, who are undergoing a comprehensive evaluation of environmental exposure, HFC and liver stiffness measurement, liver histology in those at risk of advanced fibrosis, circulating biomarkers of hepatic damage, coagulation status and early cardiovascular damage;
* To validate the causal role of HFC in the alterations of metabolism, coagulation, and early cardiovascular damage associated with NAFLD;
* To identify new inherited risk variants and microbiota profiles associated with NAFLD; to investigate the mechanism linking genetic susceptibility with liver disease and coagulation balance in in vitro models of NAFLD in hepatocytes, sinusoidal endothelial cells, and hepatic stellate cells. The investigators expect to demonstrate that the combined evaluation of genetic and novel circulating biomarkers with imaging improves the non-invasive prediction of both liver-related (leading to personalised and cost-effective surveillance of liver-related complications) and unrelated complications of NAFLD in at risk individuals, with a special focus on the role of the coagulation balance, and to pinpoint new genetic modifiers of disease progression that may be prioritized for future therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors aged between 40 and 65 years presence of clinical diagnosis of overweight or obesity (body mass index-BMI > 25 kg/m2),
* increased fasting blood glucose or T2D (fasting blood glucose ≥100mg/dl) or dyslipidemia (triglycerides≥150mg/dl, HDL<45/55 in M/F) or arterial hypertension (n = 2,452, 11.8% of the entire cohort).

Exclusion Criteria:

* subjects suffering from chronic degenerative diseases, except hypertension in good compensation and diabetes type 2 mellitus which does not require pharmacological therapy (as is already common practice for eligibility for donation of blood)
* donors aged > 65 and < 40 to avoid the introduction of bias

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
association of liver fat accumulation | up to 48 months
  At the time of enrollment, to test the association of liver fat accumulation (HFC) with liver disease and cardiovascular complications the association between HFC-genetic risk score (GRS) data will be collected on the characterization of clinical risk factors through Fibroscan measurement of liver stiffness, liver stiffness measurement (LSM) and controlled attenuation parameter (CAP), in subjects at higher metabolic risk and therefore dysteatosis. This information will be collected in the blood donor subject's management system.
the role of liver fat | up to 48 months
  The genetic risk score predicts liver fat content (HFC-GRS) can improve risk stratification of liver disease progression in NAFLD and how new common and rare genetic variants contribute to susceptibility to NAFLD. The same data also highlighted a possible new non-invasive circulating biomarker associated with liver fat and lipotoxicity (interleukin-32).
  So the evaluation of complete genetic risk scores (GRS) can be used to stratify the risk of liver-related complications and to select the best pharmacological therapy.
  Technological advances that enable the interrogation of the entire human genome, combined with the exploitation of bioinformatics systems approaches, are proving promising for providing patients and clinicians with unique health information from the molecular, cellular to multi-organ levels.
  By taking advantage of these new technologies, we assessed the role of liver fat (HFC) in coagulation alterations and influence cardiovascular risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT06566105/Prot_SAP_000.pdf